CLINICAL TRIAL: NCT02400515
Title: Influence of Regular Exercise and Detraining on Metabolic and Emotional Parameters in Diabetic and Hypertensive Individuals
Brief Title: Influence of Regular Exercise and Detraining on Metabolic and Emotional Parameters in Diabetic Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Andrea Sanches, Ms., University of Campinas, Brazil
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 030/2007
Record Dates: First submitted 2015-03-05; First posted 2015-03-27 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Exercise; Exercise Therapy; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Moderate Exercise (Other): Aerobic physical exercise was applied during 3 months, 3x/week on women with type 2 diabetic. The evaluation occurred before and after exercise in the same (and only) group, considering that this is a quasi-experimental study.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — This is a quasi-experimental study and the same group was evaluated before and after the exercise.

SUMMARY:
This quasi-experimental study aim to evaluate the effect of moderate aerobic exercise on glucose and lipid metabolism as well as the scales of anxiety and depression and levels of salivary cortisol in women with type 2 diabetes.

DETAILED DESCRIPTION:
This quasi-experimental study aim to performed a 12-week training program (3 times/week, 60 minutes per session) which consisted of a supervised moderate aerobic exercise previously determined (50% to 70% of maximal Heart Rate) in women with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* having normal physical examinations,
* no participation in regular, moderate or intensive exercise for at least 6 months before the study and
* not be following a diet

Exclusion Criteria:

* the use of insulin and beta-blocker medications and
* the functional inability to perform exercise

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-08; Primary Completion 2008-03 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Glucose levels | 3 months
  After practicing the exercise for 3 months, patients were submitted to a new collection of blood for Glucose test.

SECONDARY OUTCOMES:
Systolic and Diastolic blood pressure | 3 months
  Change in Systolic and Diastolic blood pressure were evaluated before and after physical exercise, during 3 months.
Heart Rate measurement | 3 months
  Change in heart rate was evaluated before, during and after physical exercise, during 3 months.
Glycated hemoglobin levels | 3 months
  After practicing the exercise for 3 months, patients were submitted to a new collection of blood for Glycated hemoglobin test.
Proteinuria levels | 3 months
  After practicing the exercise for 3 months, patients were submitted to a new collection of blood for proteinuria test.
Triglycerides levels | 3 months
  After practicing the exercise for 3 months, patients were submitted to a new collection of blood for triglycerides test.
High Density Level (HDL) Cholesterol levels | 3 months
  After practicing the exercise for 3 months, patients were submitted to a new collection of blood for High Density Level Cholesterol test.
Low Density Level (LDL) Cholesterol levels | 3 months
  After practicing the exercise for 3 months, patients were submitted to a new collection of blood for Low Density Level Cholesterol test.

OTHER OUTCOMES:
Salivary cortisol | 3 months
  After practicing the exercise for 3 months, patients were submitted to a new saliva collection for the salivary cortisol measure.
Hospital Anxiety and Depression scale (HADS) | 3 months
  After 3 months of the physical exercise, the HADS was evaluated.